CLINICAL TRIAL: NCT01720615
Title: Detection of Consciousness by EEG and Auditory Evoked Potentials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Gerhard Schneider, Dr. med., Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Anesthesia; Electroencephalography/ Drug Effect
Keywords: EEG; AEP; Propofol; Sevoflurane; Remifentanil; General anesthesia
MeSH Terms: interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol or Sevoflurane (No Intervention): General anesthesia
  Interventions: Drug: Propofol / Remifentanil; Drug: Sevoflurane / Remifentanil

INTERVENTIONS:
Drug: Propofol / Remifentanil — General anesthesia: Loss of consciousness and standard clinical practice
Drug: Sevoflurane / Remifentanil — General anesthesia: Loss of consciousness and standard clinical practice

SUMMARY:
The objective of the present investigation is to analyze EEG and auditory evoked potentials at the transition from consciousness to unconsciousness and vice versa. A set of electroencephalographic and auditory evoked potential parameters should be identified that allows separation of consciousness from unconsciousness (reflected by responsiveness/unresponsiveness to command). The study is based on data of 80 patients undergoing general anesthesia with remifentanil and either sevoflurane or propofol.

DETAILED DESCRIPTION:
During the past years, monitoring of anesthetic effects on the main target of anesthesia, the brain, has gained increasing attention. Monitoring of the spontaneous electroencephalogram (EEG) and of auditory evoked potentials (AEP) has been suggested. Even if EEG and AEP reflect effects of anesthetic drugs, a visual interpretation is not expedient. As a consequence, several processing methods have been suggested that reduce the electroencephalogram to a numerical value. In the current study, a set of EEG- and AEP parameters based on different analysis methods is tested with respect to the parameters ability in separating consciousness (reflected by responsiveness to command) from unconsciousness at the transition between these stages. Therefore data of 80 unpremedicated patients undergoing general anesthesia with remifentanil and either sevoflurane or propofol is used. The study period is from induction of anesthesia until patients follow command after surgery and includes a reduction of the hypnotic agent after tracheal intubation until patients follow command. The isolated forearm technique is applied before muscle relaxants are given to maintain the ability to squeeze hand to command.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-2
* Adult patients

Exclusion Criteria:

* Patients with contraindications to the study drugs
* psychiatric or neurologic disease
* drug abuse or medication known to affect the central nervous system
* pregnancy
* indication for rapid sequence induction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-01; Primary Completion 2001-11 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Changes in EEG- and AEP-parameters during loss- and return of consciousness | 1 day

SECONDARY OUTCOMES:
Impact of muscle activity on EEG- and AEP-parameters | 1 day
Influence of anesthetics on EEG- and AEP-parameters | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard F Kochs, MD, Study Chair — Klinikum rechts der Isar Technische Universität München
Locations (1):
- Technische Universität München, Klinikum rechts der Isar, Department of Anesthesiology, Munich, Bavaria, Germany